CLINICAL TRIAL: NCT00920439
Title: An Open-label Study to Assess the Safety and Reactogenicity of GlaxoSmithKline Biologicals' Inactivated Poliomyelitis Vaccine Poliorix Administered as a Booster Dose at 18-24 Months of Age in Healthy Toddlers in China.
Brief Title: Safety and Reactogenicity of GlaxoSmithKline (GSK) Biologicals' IPV Vaccine (PoliorixTM) in Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 112683
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-05

CONDITIONS: Poliomyelitis
Keywords: Poliomyelitis Vaccines; IPV
MeSH Terms: conditions — Poliomyelitis

ARMS (1):
- POLIORIX GROUP (Experimental): Healthy male or female subjects between, and including, 18 and 24 months of age, received a single booster dose of Poliorix™ vaccine that was administrated into the upper right thigh by intramuscular injection (IM).
  Interventions: Biological: PoliorixTM

INTERVENTIONS:
Biological: PoliorixTM — Single dose, intramuscular administration.

SUMMARY:
The study will evaluate the safety and reactogenicity of PoliorixTM given as a single booster dose to Chinese children at 18-24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female toddler between, and including, 18 and 24 months of age at the time of the booster vaccination.
* Subjects who received three doses of OPV as primary vaccination in the first year of life as per Chinese recommendations.
* Subjects who the investigator believes that their parents/ guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccination
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination, or planned administration during the study period, with exception of DTP and/or Hib vaccine(s).
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster vaccination, or planned administration during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Previous booster vaccination against poliomyelitis since the end of the primary vaccination series.
* History of poliomyelitis disease.
* History of seizures or progressive neurological disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Major congenital defects or serious chronic illness.

The following condition is temporary or self-limiting and a subject may be vaccinated once the condition has resolved and no other exclusion criteria are met:

• Current febrile illness or axillary temperature > 37.0 ºC or other moderate to severe illness within 24 hours of study vaccine administration.

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2009-08-03 (Actual); Study Completion 2009-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wuzhou, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Li R, Li CG, Li Y, Liu Y, Zhao H, Chen X, Kuriyakose S, Van Der Meeren O, Hardt K, Hezareh M, Roy-Ghanta S. Primary and booster vaccination with an inactivated poliovirus vaccine (IPV) is immunogenic and well-tolerated in infants and toddlers in China. Vaccine. 2016 Mar 14;34(12):1436-43. doi: 10.1016/j.vaccine.2016.02.010. Epub 2016 Feb 9. PMID 26873055
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 112683 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112683 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112683 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112683 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112683 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112683 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 26 subjects enrolled in the study, one did not receive any vaccination.
Groups:
- Poliorix Group: Healthy male or female subjects between, and including, 18 and 24 months of age, received a single booster dose of Poliorix vaccine that was administrated into the upper right thigh by intramuscular injection (IM).
Period: Overall Study
Arm/Group | Poliorix Group
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Poliorix Group
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Months] | 20.3 (1.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = all reports of the specified symptom irrespective of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with documented administration of the study vaccine.
Measure: Number; unit: Subjects
Arm/Group | Poliorix Group
Number analyzed (Participants) | 25
Subjects
  Any Pain | 4
  Grade 3 Pain | 0
  Any Redness | 5
  Grade 3 Redness | 0
  Any Swelling | 3
  Grade 3 Swelling | 0

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were temperature [defined as axillary temperature equal to or above (≥) 37.1 degrees Celsius (°C)], drowsiness, irritability and loss of appetite. Any = all reports of the specified symptom irrespective of intensity grade and relationship to vaccination. Grade 3 drowsiness= drowsiness that prevented normal activity. Grade 3 irritability= crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite= subject did not eat at all. Grade 3 fever = fever above (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Poliorix Group
Number analyzed (Participants) | 25
Subjects
  Any Drowsiness | 3
  Grade 3 Drowsiness | 0
  Related Drowsiness | 3
  Any Irritability | 5
  Grade 3 Irritability | 0
  Related Irritability | 3
  Any Loss of appetite | 3
  Grade 3 Loss of appetite | 0
  Related Loss of appetite | 2
  Any Temperature | 6
  Grade 3 Temperature | 0
  Related Temperature | 5

3. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Poliorix Group
Number analyzed (Participants) | 25
Subjects
  Any AE(s) | 10
  Grade 3 AE(s) | 0
  Related AE(s) | 0

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 to Month 1)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Poliorix Group
Number analyzed (Participants) | 25
Subjects | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4-day (Days 0-3) post-vaccination period. Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period. SAEs: during the entire study period (from Day 0 up to Month 1).
Arm/Group | Poliorix Group
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 14/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poliorix Group (N=25)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5)
Irritability (Psychiatric disorders) | 5 (5)
Nasopharyngitis (Infections and infestations) | 3 (4)
Pain (General disorders) | 4 (4)
Pyrexia (General disorders) | 7 (10)
Somnolence (Nervous system disorders) | 3 (3)
Swelling (General disorders) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.